CLINICAL TRIAL: NCT00548834
Title: Efficacy and Safety of CDP870 400 mg Subcutaneously Versus Placebo in the Treatment of the Signs and Symptoms of Patients With Rheumatoid Arthritis Who Have Previously Failed at Least One DMARD
Brief Title: Efficacy and Safety of CDP870 Versus Placebo in the Treatment of the Signs and Symptoms of Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C87011
Record Dates: First submitted 2007-10-15; First posted 2007-10-24 (Estimated); Last update posted 2013-09-04 (Estimated); Status verified 2010-02

CONDITIONS: Rheumatoid Arthritis
Keywords: CDP870; Certolizumab Pegol
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Certolizumab Pegol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: CDP870

SUMMARY:
The purpose of this study was to confirm and extend the data from previous studies and to demonstrate the efficacy (in terms of signs and symptoms) and safety of monotherapy with CDP870 administered SC every 4 weeks compared to placebo in patients with active RA who had failed at least one DMARD.

ELIGIBILITY:
Inclusion Criteria:

* male/female, 18-75 years old, inclusive
* diagnosis of adult-onset RA
* had active disease
* had received methotrexate
* on a stable dose of folic acid

Exclusion Criteria:

* contraindication for methotrexate or anti-TNF

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2003-06; Primary Completion 2004-07 (Actual); Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
American College of Rheumatology (ACR)-20 responder rate at Week 24 | 24 weeks

SECONDARY OUTCOMES:
safety and tolerability every 4 weeks | Every 4 weeks
effect of CDP870 on health outcomes measures | 24 weeks
systemic exposures and immunogenic profile of CDP870 | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — UCB Pharma

REFERENCES:
- [Result] Fleischmann R, Vencovsky J, van Vollenhoven RF, Borenstein D, Box J, Coteur G, Goel N, Brezinschek HP, Innes A, Strand V. Efficacy and safety of certolizumab pegol monotherapy every 4 weeks in patients with rheumatoid arthritis failing previous disease-modifying antirheumatic therapy: the FAST4WARD study. Ann Rheum Dis. 2009 Jun;68(6):805-11. doi: 10.1136/ard.2008.099291. Epub 2008 Nov 17. PMID 19015206